CLINICAL TRIAL: NCT03044886
Title: Effects of Vitamin D on Chronic Periodontitis
Brief Title: Effects of Vitamin D on Moderate to Severe Periodontitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Chao Yang Hospital (Other)
Responsible Party: Principal Investigator, Zuo Min Wang, Dean of Stomatology Department, Beijing Chao-Yang Hospital, Beijing Chao Yang Hospital
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: BeijingCYH1
Record Dates: First submitted 2017-01-17; First posted 2017-02-07 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2019-02-18 (Actual); Status verified 2019-02

CONDITIONS: Chronic Peritonitis
Keywords: Vitamin D
MeSH Terms: interventions — Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (3):
- 2000IU/day (Experimental): Subjects took 2000IU vitamin D per day
  Interventions: Dietary Supplement: vitamin D
- 1000IU/day (Experimental): Subjects took 1000IU vitamin D per day
  Interventions: Dietary Supplement: vitamin D
- Placebo (Placebo Comparator): Subjects took placebo
  Interventions: Dietary Supplement: vitamin D

INTERVENTIONS:
Dietary Supplement: vitamin D — Subjects took vitamin D or placebo

SUMMARY:
The object of the study was to evaluate the direct effect of high dose vitamin D supplementation on chronic periodontitis, and suggest the recommended dose for clinic use.

DETAILED DESCRIPTION:
Periodontitis is a chronic inflammatory disease characterized by periodontal tissues inflammation and alveolar bone loss. Vitamin D is involved in stimulating osteoblasts to enable normal bone growth and preservation, also the regulation of cellular proliferation, differentiation, innate immune response and anti-inflammatory effect.Previous studies have reported the association of vitamin D levels and gingivitis and periodontitis. This study was designed as a randomized controlled trial to evaluate the effect of vitamin D supplementation on chronic periodontitis.

The study was divided into two phases. Recruitment including baseline clinical measurements was obtained and standard periodontal treatments were performed in Phase One. The randomization and intervention of vitamin D were performed in Phase Two. The 323 subjects were randomly divided into 3 groups (n=105,110,108) to receive a supplement kit containing 90 capsules of 2000 IU vitamin D, 1000 IU vitamin D, or placebo capsule for 3 months. After intervention, all the subjects were followed up after 3 months and received standard periodontal examination, including attachment loss (AL), probing depth (PD), bleeding index (BI), and panoramic radiographs were taken to evaluate alveolar crest height (ACH).

ELIGIBILITY:
Inclusion Criteria:

1. Age from 30 years old to 70 years old
2. More than 20 teeth remaining in the mouth
3. Clinical diagnosis of moderate to severe periodontitis
4. Not receiving periodontal treatment within 6 months
5. Not taking antibiotic drugs within 3 months.

Exclusion Criteria:

1. Diabetes, thyroid and parathyroid endocrine associated diseases
2. Severe systemic diseases, such as cancer
3. Taking vitamin D and / or calcium drugs during observation
4. Taking aspirin, non-steroidal anti-inflammatory drugs, and steroids
5. Pregnant or prepare to pregnant within one year
6. Have been suffering from hypercalcemia, malabsorption syndrome.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2013-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zuomin Wang, Doctor, Principal Investigator — Dean of Stomatology Department

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Started | 120 | 120 | 120
Completed | 105 | 110 | 108
Not Completed | 15 | 10 | 12
Not completed — Lost to Follow-up | 15 | 10 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo | Total
Number analyzed (Participants) | 120 | 120 | 120 | 360
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 103 | 110 | 107 | 320
  >=65 years | 17 | 10 | 13 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 49 (5.4) | 51 (6.3) | 53 (5.2) | 51 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 59 | 62 | 57 | 178
  Male | 61 | 58 | 63 | 182
Region of Enrollment [Number; unit: participants]
  China | 120 | 120 | 120 | 360

OUTCOME MEASURES:

1. Primary Outcome: Attachment Loss (AL)
Description: Examination of AL was performed with Williams probe, included six sites of each tooth: mesial buccal, buccal, distal buccal, mesial lingual, lingual and distal lingual. The outcome was the mean value of all the sites of all subjects.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 4.7 (1.1) | 4.8 (0.9) | 4.8 (0.9)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.576, ANOVA

2. Primary Outcome: Attachment Loss (AL)
Description: as for outcome 1
Time Frame: 3 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 3.5 (0.7) | 3.6 (0.7) | 3.6 (0.6)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; Test type: Superiority; p = 0.489, ANOVA

3. Primary Outcome: Attachment Loss (AL)
Description: as for outcome 1
Time Frame: 6 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 3.4 (0.6) | 3.3 (0.6) | 3.3 (0.7)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; Test type: Superiority; p = 0.042, ANOVA
Statistical Analysis 2: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine changes from 3 month to 6 month of all groups; Test type: Superiority; p = 0.041, ANOVA

4. Secondary Outcome: Probing Depth (PD)
Description: Examination of PD was performed with Williams probe, included six sites of each tooth: mesial buccal, buccal, distal buccal, mesial lingual, lingual and distal lingual. The outcome was the mean value of all the sites of all subjects.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 3.6 (0.8) | 3.7 (0.8) | 3.6 (0.7)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.710, ANCOVA

5. Secondary Outcome: Probing Depth (PD)
Description: as for outcome 4
Time Frame: 3 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 2.5 (0.5) | 2.6 (0.4) | 2.6 (0.5)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; Test type: Superiority; p = 0.340, ANOVA

6. Secondary Outcome: Probing Depth (PD)
Description: as for outcome 4
Time Frame: 6 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 2.4 (0.5) | 2.5 (0.4) | 2.5 (0.4)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; Test type: Superiority; p = 0.048, ANOVA
Statistical Analysis 2: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.038, ANOVA

7. Secondary Outcome: Alveolar Crest Height (ACH)
Description: Panoramic radiographs were taken to evaluate alveolar crest height (ACH) with measuring software (i-Dixel, One Volume Viewer, version 6.00, J. MORITA MFG. CORP. Japan). The alveolar crest height is defined as the mean of the two-dimensional vertical distance between mesial and distal alveolar crest to apical point.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 7.7 (2.3) | 7.7 (2.2) | 7.8 (2.4)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.521, ANOVA

8. Secondary Outcome: Alveolar Crest Height (ACH)
Description: as for outcome 7
Time Frame: 3 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 7.7 (2.1) | 7.6 (2.3) | 7.7 (2.1)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.742, ANOVA

9. Secondary Outcome: Alveolar Crest Height (ACH)
Description: as for outcome 7
Time Frame: 6 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
mm | 7.7 (2.3) | 7.7 (2.2) | 7.7 (2.0)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p < 0.05, ANOVA
Statistical Analysis 2: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.073, ANOVA

10. Secondary Outcome: Bleeding Index (BI)
Description: Examination of BI was performed with Williams probe, explored under the gingival margin about 1mm, and bleeding was observed after 30 seconds. BI was scored on a 0-5 scale, higher scores mean a worse outcome.
Time Frame: at baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
score on a scale | 3.5 (1.1) | 3.2 (1.3) | 3.8 (1.2)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.348, ANOVA

11. Secondary Outcome: Bleeding Index (BI)
Description: as for outcome 10
Time Frame: 3 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
score on a scale | 1.5 (0.8) | 1.7 (0.6) | 1.6 (0.8)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.685, ANOVA

12. Secondary Outcome: Bleeding Index (BI)
Description: as for outcome 10
Time Frame: 6 months after periodontal treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
Number analyzed (Participants) | 105 | 110 | 108
score on a scale | 0.9 (0.3) | 1.2 (0.7) | 1.1 (0.6)
Statistical Analysis 1: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; One-way analysis of variance (ANOVA) and Neuman-Keuel test were carried out to determine difference between groups; Test type: Superiority; p = 0.075, ANOVA
Statistical Analysis 2: Comparison: 2000IU/Day vs 1000IU/Day vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority; p = 0.083, ANOVA

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 6 months
Arm/Group | 2000IU/Day | 1000IU/Day | Placebo
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/120
Other Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 0/120

LIMITATIONS AND CAVEATS:
The observation time was short. Mechanical periodontal therapy might be too close in time to the vitamin D treatment. Did not adjust for possible confounding factors (e.g., dietary vitamin D) . The study was performed at one single center.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes